CLINICAL TRIAL: NCT04904250
Title: SpiderFX Versus Emboshield Nav6 Distal Protection on Cerebral Microembolization in Vulnerable Plaque During Carotid Artery Stenting
Brief Title: Spider Versus Emboshield Distal Protection on Cerebral Microembolization During Vulnerable Plaque in Carotid Artery Stenting
Acronym: CASH-ES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CASH-ES
Record Dates: First submitted 2021-04-30; First posted 2021-05-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Carotid Stenosis; Carotid Artery Stent
Keywords: stroke; carotid stenosis; carotid artery stenting
MeSH Terms: conditions — Stroke; Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emboshield NAV6 (Experimental): using Emboshield NAV6 distal embolism protection device during CAS
  Interventions: Device: Emboshield
- SpiderFX (Active Comparator): using SpiderFX distal protection device during CAS
  Interventions: Device: Spider

INTERVENTIONS:
Device: Emboshield — a distall occlusion Emboshield NAV6 will be used as the embolism protection device during CAS
  Other Names: Emboshield NAV6 (Abbott vascular, Santa Clara, CA, USA)
  Arms: Emboshield NAV6
Device: Spider — a distal SpiderFX will be used as the embolism protection device during CAS
  Other Names: SpiderFX (Medtronic, Minneapolis, Minnesota, USA)
  Arms: SpiderFX

SUMMARY:
A single center, prospective, outcome-assessor-blinded, randomized controlled trial study (CASH-ES) is designed to compare the efficiency of two different distal embolism protection devices (SpiderFX and Emboshield NAV6) in during CAS procedure of patients with vulnerable plaque.

DETAILED DESCRIPTION:
CAS is an alternative to CEA for treating carotid stenosis with a similar efficacy in preventing future stroke. High-intensity signal in the plaque on the TOF-MRA is associated to a high risk of cerebral embolism during stenting. The evidence of protection selection in such patients was limited. A single center, prospective, outcome- assessor-blinded, randomized controlled trial study (CASH-ES) is designed to compare the efficiency of two distal embolism protection devices (SpiderFX and Emboshield NAV6) during CAS procedure of patients with vulnerable plaque. Asymptomatic patients with internal carotid artery stenosis ≥ 70% (NASCET) and symptomatic patients with a stenosis ≥ 50% who is over 70 years old, diagnostic of vulnerable plaque on ultrasound or have a high-intensity signal in the relevant plaques on TOF-MRA will be included. Patients are randomized in two balanced groups (1:1) to receive CAS with either distal (Spider FX) or distal (Emboshield NAV6) protection. The primary endpoint is the incidence of new cerebral ipsilateral ischemic lesions on the DW-MRI within 7-days post operation. Secondary endpoints include the number, size, location of new cerebral ischemic lesions on the DW-MRI, the counts of MES during TCCD monitoring during procedure, procedural complications, stroke, myocardial infarction, and death within 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age and older.
2. Symptomatic patients with internal carotid artery stenosis≥50% on angiography, or asymptomatic patients with internal carotid artery stenosis≥70% on angiography.
3. Anatomic characteristics of the lesions that made it possible to use either type of distal embolism protective device (Emboshield or Spider).
4. The lesion was located in the internal carotid artery (ICA) or the bifurcation of the carotid artery.
5. Only one WALLSTENT is expected to treat target lesions.
6. Tolerance to aspirin/clopidogrel/heparin and other drug therapy.
7. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Medical Ethics Committee, Institutional Review Board, or Human Research Ethics Committee.
8. High-intensity Signal in the relevant plaques on the TOF-MRA.

Exclusion Criteria:

1. Extensive ipsilateral or disabling stroke(mRS≥2) or cerebrovascular events occurred within 1 month combined with neurological defects.
2. Myocardial infarction occurred within 72 hours or TIA within 48 hours.
3. Atrial fibrillation (chronic or paroxysmal) is not treated with anticoagulation.
4. Ipsilateral intracranial artery stenosis with a history of stenting.
5. CABG or vascular surgery in the 30-day period before the procedure.
6. Acute coronary syndrome in the 30-day period before the procedure.
7. Life span within 12 months.
8. Patient has a history of bleeding diathesis within 1 month or coagulopathy or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated.
9. Intolerance or allergic reaction to a study medication without a suitable management alternative.
10. The femoral artery condition is not good enough to enter the guidewire or the sound window is not good enough to conduct intraoperative TCD monitoring of the patient.
11. Unfavorable femoral artery anatomy for endovascular intervention or unfavorable acoustic window for intraoperative TCD monitoring.
12. With Intracranial tumor and is not considered suitable for inclusion or could not complete the MRI examination.
13. WBC<3*109/L, PLT<50*109/L or >700*109/L.
14. Pregnant or lactating female patient.
15. DSA indicated the target vessel occlusion; The tandem lesions could not be covered by one stent; The target vessel was seriously tortuous or the internal carotid artery was not suitable for WallStent; The aortic arch has severe calcification or tortuosity involving the common carotid artery or brachial trunk; Combined with cerebral AVM or cerebral aneurysms which need treatment; Carotid artery stenosis not caused by atherosclerosis, but arteritis, arterial dissection, congenital malformation of blood vessels, or severe vascular lesions after radiotherapy, etc..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-08-27 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral new ischemic lesions on DWI | Within 7 days post-operation
  The incidence of ipsilateral new ischemic lesions on DWI after CAS

SECONDARY OUTCOMES:
major stroke | within 7 days post-operation
  the incidence of major stroke after CAS, defined as new onset of neurological symptoms causing an increase of NIHSS ≥ 4 or worsening of existing focal neurological deficit lasting ≥ 24 hours
myocardial infarction | within 7 days post-operation
  the incidence of myocardial infarction after CAS, defined as new onset of chest discomfort or cardiac stroke or heart failure with a rise and/or fall of cardiac biomarkers and ECG abnormalities
death | within 7 days post-operation
  In-hospital mortality
Any hemorrhage, acute kidney injury and other procedure-related complications | within 7 days post-operation
  including major/minor hemorrhage, acute kidney injury, etc.
The number of new cerebral ischemic lesions on DW-MRI | within 7 days post-operation
  The number of new cerebral ischemic lesions on DW-MRI
The size of new cerebral ischemic lesions on DW-MRI | within 7 days post-operation
  The size of new cerebral ischemic lesions on DW-MRI
The location of new cerebral ischemic lesions on DW-MRI | within 7 days post-operation
  The location of new cerebral ischemic lesions on DW-MRI
MES counting during CAS | during CAS procedure
  TCD monitoring of MES counting during CAS

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, PhD, Principal Investigator — Department of Interventional Neuroradiology, Department of Neurosurgery, International Neuroscience Institute (China-INI), Xuanwu Hospital, Capital Medical University
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No